CLINICAL TRIAL: NCT03248713
Title: Glucocorticoid Antagonist Treatment for Tobacco Use Disorder
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: MS053
Record Dates: First submitted 2017-08-04; First posted 2017-08-14 (Actual); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Mifepristone; Sugars

STUDY DESIGN:
Intervention Model Description: The primary analyses will use linear mixed models (LMMs). LMMs can handle continuous and dichotomous outcomes, as well as missing data. Analyses will include baseline (pre-treatment) measures of these variables as covariates and other baseline variables where appropriate.
Who Masked: Participant, Investigator
Masking Description: This is a double blind randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mifepristone (Active Comparator): Mifepristone 600 mg/day in 2 tablets
  Interventions: Drug: Placebo
- Placebo (Placebo Comparator): matching placebo in 2 tablets
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Mifepristone 600mg 2 tablets will be compared to the placebo
  Other Names: korlym, mifeprex
  Arms: Placebo
Drug: Placebo — Placebo sugar 2 tablets will be compared to mifepristone
  Other Names: sugar pill
  Arms: Mifepristone

SUMMARY:
The purpose of this protocol is to examine whether mifepristone, a medication with glucocorticoid receptor antagonist activity, may be a potential treatment for Tobacco Use Disorder (TUD). Mifepristone has already shown promise as a potential treatment for PTSD (1) and alcohol use disorder (AUD) (2), but no previous studies have examined the therapeutic potential of mifepristone for TUD. This will be a double-blind, placebo-controlled study on the effects of a 7-day treatment with 600 mg mifepristone, or placebo, on cognitive function, tobacco withdrawal severity, and smoking behavior.

DETAILED DESCRIPTION:
This will be a double-blind, placebo-controlled study that tests the effects of a 7-day treatment with 600 mg mifepristone, or placebo, on cognitive function, tobacco withdrawal severity and smoking behavior. Once the intake and physical examination is completed and eligibility is determined, subjects will participate in a baseline session to become familiar with the study procedures and to assess baseline measures of withdrawal, smoking urges, pain sensitivity, and cognitive performance. Subjects will be asked to refrain from consuming alcoholic beverages and drugs during their study participation. This will be verified by urine drug screening and breathalyzer before the session and during outpatient visits. If results indicate non-compliance with these study procedures, subjects will be discharged from the study.

Participants will be assessed for compliance with medication treatment, withdrawal severity, recent smoking behavior, and cognitive function during treatment visits on Days 1 and 4. On Day 7, following overnight abstinence from smoking, participants will attend a test session that models relapse to smoking. During this session, subjects will have the option to smoke, or to delay smoking in exchange for monetary compensation (45). To examine if mifepristone's proposed therapeutic effects last beyond the treatment duration (as observed in previous studies), there will be 1-week and 1-month follow-up assessments on smoking behavior, urges to smoke, endocrine biomarkers, and cognitive function.

Participants in each group will complete the laboratory-based, delayed smoking procedure in a designated, negative pressure room in Bldg. 36 of the West Haven VA just after assessing pain sensitivity with the cPT. This sequence allows the cPT to assess pain sensitivity, a potential biomarker of relapse behavior, and to also be used as a mild stressor prior to participation in the smoking relapse model. Participants will be instructed to abstain from smoking after 10 pm the night before Test Sessions. Abstinence will be confirmed the morning of the session by measuring a breath CO level of < 8 ppm.

ELIGIBILITY:
Inclusion Criteria:

* Male smokers aged 18 to 55 years;
* History of smoking at least 5 cigarettes daily for the past 12 months;
* In good health as verified by medical history, screening examination, and -screening laboratory tests

Exclusion Criteria:

* History of mifepristone allergy;
* Requirement of any form of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics) and recent psychiatric history (in the past 6 months);
* Medical illnesses including diabetes, cardiovascular, renal, endocrine, or hepatic disorders;
* Prolonged QTc interval >450 msec;
* History of adrenal insufficiency or a morning plasma cortisol level less than 5 mcg/dl at screening;
* Hypokalemia at screening (defined as potassium level < 3.5 mEq/L);
* Current use of clinically significant CYP 3A4 substrates including, simvastatin, lovastatin, cyclosporine, ergotamines, fentanyl, pimozide, quinidine, sirolimus, tacrolimus, triazolam, midazolam.
* use of rifapentin, phenobarbital, phenytoin, carbamazepine, and St. John's Wort.
* Current use of strong 3A4 inhibitors including ketoconazole, itraconazole, nefazodone, ritonavir, nelfinavir, indinavir, atazanavir, amprenavir, fosamprenivir, boceprevir, clarithromycin, conivaptan, lopinavir, mibefradil, posaconazole, saquinavir, telaprevir, telithromycin, voriconazole.
* Treatment with systemic corticosteroids
* Current use of clinically significant CYP 3A inducers (e.g., rifampin, rifabutin);
* Abuse of alcohol or any other illicit or prescription drugs;
* Inability to tolerate cold exposure due to conditions such as peripheral -vascular disease or Raynaud's phenomenon;
* Inability to fulfill all scheduled visits and examination procedures throughout the study period.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male smokers
Enrollment: 8 (Actual)
Dates: Start 2017-11-29 (Actual); Primary Completion 2019-05-20 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Minnesota Nicotine Withdrawal Symptom Checklist (M-NWSC) | one week
  Smokers will be asked to rate several nicotine withdrawal symptoms on a 100 mm scale, from "not at all" to "extremely."

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D.,Ph.D., Principal Investigator — Yale University
Locations (1):
- Veterans Affairs Hospital, West Haven, Connecticut, United States